CLINICAL TRIAL: NCT06846697
Title: Comparison of Hatha Yoga and Reformer Pilates Exercises on Posture, Pain, Balance, Quality of Life, Body Image and Composition and Respiratory Functions in Individuals With Hyperkyphosis
Brief Title: Effects of Hatha Yoga and Reformer Pilates on Hyperkyphosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Betül Taşpınar, Prof. Dr., Izmir Democracy University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hyperkyphosis-35
Record Dates: First submitted 2025-02-05; First posted 2025-02-26 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Hyperkyphosis
Keywords: Hatha Yoga; Reformer Pilates
MeSH Terms: conditions — Kyphosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Other): This group will be given a home programme. They will be asked to do the exercises regularly and fulfil the recommendations given and will be asked to come to the control at the end of 8 weeks. During this period, individuals will be followed up weekly by telephone.
  Interventions: Other: Home-based Exercise
- Hatha Yoga Group (Experimental): Participants in this group, who will also be given a home programme, will participate in Hatha yoga exercises 3 times a week for a total of 8 weeks with a session duration of 45 minutes, accompanied by a physiotherapist with a yoga instructor certificate. In this group, Hatha yoga exercises will be applied by focusing on postural control and respiration during exercise.
  Interventions: Other: Home-based Exercise; Other: Hatha Yoga Group
- Reformer Pilates Group (Experimental): In this group, which will be given a home programme, participants will perform the exercises 3 times a week for a total of 8 weeks with a session duration of 45 minutes, accompanied by a physiotherapist with a pilates instructor certificate.In this group, which will be given a home programme, participants will perform the exercises 3 times a week for a total of 8 weeks with a session duration of 45 minutes, accompanied by a physiotherapist with a pilates instructor certificate. In this group, reformer pilates exercises will be applied by focusing on postural control during exercise.
  Interventions: Other: Home-based Exercise; Other: Reformer Pilates Group

INTERVENTIONS:
Other: Home-based Exercise — The subjects in this group will be given the exercises included in the Physical Activity guideline of the Ministry of Health as a home programme.
  Other Names: HBE
Other: Hatha Yoga Group — The sessions will begin with the classic sun salutation series (Suryanamaskar) consisting of 12 basic poses of yoga. The sun salutation series will be used as a warm-up for 10 minutes. After warming up, postures aimed at stretching the front group muscles of the body and strengthening the back group muscles will be preferred. In the cooling phase, the session will be ended by relaxing with Savasana pose for 10 minutes.
  Other Names: HYG
  Arms: Hatha Yoga Group
Other: Reformer Pilates Group — Exercise sessions will start with the foot series and the starting position on the back will be preferred. This series, which is progressed by maintaining the body composition, is considered as a warm-up exercise of the body. Then, the body is continued with exercise series targeting the thoracic region and core region.
  Other Names: RPG
  Arms: Reformer Pilates Group

SUMMARY:
The vertebral column is an S-shaped structure that carries the body weight and transmits it to the feet. Kyphosis, a natural curvature of the spine, can increase with poor posture and muscle weakness, leading to postural kyphosis. This condition results in forward head positioning, rounded shoulders, and scapular winging, causing back pain, poor posture, balance issues, and respiratory difficulties. With technological advances, poor posture habits have become more common, especially in adolescents. Kyphosis can also affect balance, walking speed, and increase the risk of falls in older adults. Exercises like Hatha yoga and reformer Pilates are effective methods for improving posture, muscle strength, and quality of life. The aim of this study is to compare the effects of Hatha yoga and reformer Pilates exercises on posture, pain, balance, quality of life, body image, and respiratory function in individuals with hyperkyphosis.

DETAILED DESCRIPTION:
The vertebral column is an S-shaped structure that supports the weight of the upper extremities, head, and neck, transmitting this load to the pelvis and ultimately to the feet. It consists of 34-35 vertebrae, including cervical, thoracic, lumbar, sacral, and coccygeal vertebrae. The cervical and lumbar regions form concave curves (lordosis), while the thoracic and sacral-coccygeal regions form convex curves (kyphosis). The arrangement of the vertebral column in the sagittal plane enables individuals to perform activities with minimal energy expenditure. Kyphosis is the angular and physiological posture formed by the spine and surrounding muscles, which includes the vertebrae and intervertebral discs.This angle is commonly assessed using the Cobb angle in lateral radiographs, with the angle between the lines drawn perpendicular to the 4th-5th thoracic vertebrae and the 12th thoracic vertebrae being measured. Postural kyphosis is defined as an increase in existing spinal curvature due to muscle weakness and poor posture, and it is considered a more flexible deformity compared to other types of kyphosis.The mechanical changes associated with postural kyphosis can impact various functions. The head in kyphotic posture moves forward, altering cervical alignment. This causes the cervical vertebrae to shift anteriorly, leading to compensatory rounding of the shoulders and scapular winging.Factors such as prolonged sitting at desks, poor posture, inadequate furniture, physical inactivity, and heavy school bags contribute to increased muscle spasms and weakened soft tissues, aggravating kyphotic posture. Additionally, technological advancements, especially the widespread use of computers and smartphones, have led to poor postural habits in individuals, particularly adolescents.Rapid growth during adolescence can also cause abnormal spinal flexion, negatively affecting organ development and increasing the kyphosis angle.A study conducted in 2024 showed that corrective exercises combined with active diaphragmatic breathing led to improvements in chest pain and respiratory function in postmenopausal women after a 12-week program.Postural kyphosis is often asymptomatic, but it can result in a visible hunchback, poor posture, back and neck pain, tension, and sensitivity in the spine.In postural kyphosis, the individual can actively or passively correct the posture, but the curvature is flexible. Structural deformities in the spine do not occur. Incorrect postures increase stress on the joints, impairing their function and leading to pain and edema in the discs.Inadequate posture also strains bones, muscles, and ligaments, leading to pain and negatively impacting the position and function of internal organs.Balance refers to the ability to maintain the center of mass within the limits of a base of support during functional activities, utilizing vestibular, visual, and proprioceptive senses. It is classified into static balance, where the center of mass remains stable in a fixed position, and dynamic balance, which involves maintaining balance during movement. Literature indicates that individuals with increased kyphosis experience balance impairments, but postural kyphosis is not routinely assessed for balance.Some studies suggest that kyphosis negatively impacts physical function, balance, and mortality, while others have found no significant link between kyphosis and balance. Research has shown that kyphosis in older women is associated with slower walking speeds, increased body sway, balance issues, and higher fall rates.However, clinical exercises combined with breathing techniques have demonstrated improvements in quality of life and kyphosis angles.Postural kyphosis can impact both physical and psychological well-being, as it affects an individual's appearance. In young individuals, the normal thoracic kyphosis angle is between 20° and 40°, with angles over 45° considered hyperkyphosis.Exercise positively influences both mental and physical health. In adolescence, body image is crucial, and postural deviations often reflect emotional states, with extension positions fostering happiness and confidence, while flexion positions are associated with sadness.Respiration involves coordinated muscle activity. Although inspiration primarily occurs through diaphragmatic muscle activity, additional inspiratory muscles are engaged during deep inspiration. These muscles assist in expanding and contracting the thoracic cavity and contribute to stabilizing the thorax and abdomen.Postural changes in the body and shoulder girdle directly affect thoracic and diaphragm movements, influencing respiratory function. Restrictions in thoracic expansion or diaphragm movement, such as those caused by hyperkyphosis and scapular winging, limit respiratory capacity.Hyperkyphosis can lead to restrictive pulmonary dysfunction, similar to scoliosis, and increases the antero-posterior diameter of the thorax, reducing lung capacity.Studies have shown that hyperkyphosis is associated with decreased pulmonary function and lung volumes.Conservative treatments are the first line of management for postural kyphosis. Manual therapy techniques,postural correction exercises,postural taping,orthotics and the Schroth method are commonly used. Prevention of postural kyphosis begins in childhood with the teaching of proper posture, supporting exercises, muscle strengthening, and spinal alignment.Yoga and Pilates exercises are among the methods used to address these issues.Multidisciplinary treatment approaches are recommended in complementary therapies, addressing patients not only from a bio-psycho-social perspective but also through a bio-mental-physical-psycho-social understanding. Yoga, a mind-body exercise, is often recommended in group therapies. Originating in India over 4,000 years ago, yoga has developed over time to promote both physical strength and spiritual awareness. Various types of yoga, such as Hatha yoga, are similar to physiotherapy practices.Yoga incorporates postures (asanas), breathing exercises (pranayama), and meditation to improve flexibility, strength, and relaxation.Pilates, developed by Joseph Pilates in the 1900s, focuses on improving spinal stability, breathing control, and kinesthetic awareness, promoting both muscle relaxation and mental relaxation. Clinical Pilates is used in rehabilitation for both healthy individuals and those with various medical conditions.Research has shown that Pilates improves flexibility, reduces pain, and enhances quality of life and functional capacity.Studies also suggest that Pilates and yoga improve posture and balance in individuals with hyperkyphosis, although research comparing both approaches is limited.The aim of this study is to compare the effects of Hatha yoga and reformer Pilates exercises on posture, pain, balance, quality of life, body image, body composition, and respiratory function in individuals with hyperkyphosis.

ELIGIBILITY:
Inclusion Criteria:

* Postural hyperkyphosis
* Not receiving physiotherapy in the last 6 months

Exclusion Criteria:

* Exercise is not indicated
* Communication problems
* Having a concomitant orthopaedic disorder
* The presence of a concomitant neurological disorder
* Presence of concomitant cardiopulmonary disease
* Presence of recurrent infection
* Presence of open wound and/or incision
* Presence of other spinal conditions such as scoliosis
* Being diagnosed with kyphosis other than postural kyphosis in the classification system
* Previously undergone a related surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
New York Posture Evaluation Scale | At baseline and after 8 weeks
  The New York Posture Evaluation Scale was first published in 1958. It evaluates the body in 13 different parts in terms of posture changes that may occur. If the posture is correct, 5 points are given, 3 points if it is moderately impaired, and 1 point if it is severely impaired. The total score obtained as a result of the test varies between 13-65 points. A high score means that the posture is good.
Measurement of the degree of kyphosis with Flexicurve | At baseline and after 8 weeks
  Flexicurve will be used to determine the degree of hyperkyphosis. Flexicurve, a noninvasive method, is recommended as a practical and affordable tool for monitoring age-related spinal degenerative processes and curvature changes. One end of the Flexicurve is placed on the bony prominence of the cervical seventh (C7) vertebra and caudally along the spine to the thoracic twelfth vertebra. The mould is then removed from the spine and the shape transferred to paper. Showing the relationship between the length and width of the thorax; Values are obtained according to the formula (width / length) x 100
Determination of the distance between the occiput and the wall | At baseline and after 8 weeks
  It is a practical method widely used for screening and monitoring hyperkyphosis. The individual's back and heels should be as close to the wall as possible and the head should remain in a natural position. Hyperkyphosis is considered to be present if the occiput does not touch the wall when the back and heels are against the wall and the head is facing forwards. The degree of hyperkyphosis is assessed by measuring the distance between the occiput and the wall. The severity of hyperkyphosis is classified as mild (≤5 cm), moderate (5.1-8 cm) and severe (>8 cm).
Determination of the distance between wall C7 | At baseline and after 8 weeks
  There are also studies suggesting that it would be more appropriate to use C7 in the measurement because it is closer and adjacent to the thoracic vertebrae than the occiput. Due to the close location of C7 to the thoracic vertebrae, errors that may be encountered when the participant moves his/her head will be prevented. The measurement is performed with the back, heels and sacrum against the wall, in as upright a posture as possible and looking forwards. The distance of the spinous process of C7 perpendicular to the wall is measured using two rulers. According to the test results, the severity of hyperkyphosis is expressed in three different levels: mild (≤ 5 cm), moderate (5.1- 8 cm) and severe (> 8 cm).
Visual Analogue Scale | At baseline and after 8 weeks
  Perceived pain ranges from no pain to extreme pain. For pain intensity according to the VAS, 'no pain' is graded as 0 points and 'worst possible pain' is graded as 10 points.
Timed balance test | At baseline and after 8 weeks
  In this test, the duration of standing on one and two legs with eyes open and closed is analysed. It is a static balance test
Flamingo balance test | At baseline and after 8 weeks
  It is a test that measures the duration of static balance in seconds within a one-minute evaluation process. The tool used as an auxiliary material is fixed on the floor. The person conducting the research sits facing the person with the stopwatch. The second observer stands next to the person to help ensure the balance of the person and to see the number of errors in the instrument. One foot of the person stays in the air during this test and when this foot touches the ground or when the person drops this foot completely, the error is recorded and the stopwatch is stopped. After the balance is restored, the stopwatch is restarted and the best score is taken and recorded as the test score. If the person makes fifteen or more errors within 30 seconds after the balance is restored, the test score is reflected as 0.
Timed up and go test | At baseline and after 8 weeks
  This test requires a chair, a stopwatch and a three-metre walking space. The test starts with sitting on a chair, the individual gets up with a warning, walks 3 metres, returns and sits down. It is a test used in dynamic balance assessment.
Functional reach test | At baseline and after 8 weeks
  With the help of a tape measure mounted on the wall, the ability of the subjects to reach without losing their balance is evaluated. It is a test used in dynamic balance assessment.
Nottingham Health Profile (NHP) | At baseline and after 8 weeks
  It is used to assess quality of life. The questionnaire consists of 38 items. It evaluates six dimensions of quality of life including energy; 3 items, pain; 8 items, emotional reactions; 9 items, sleep; 5 items, social isolation; 5 items, physical activity; 8 items. Each section is scored between 0-100, '0' indicates the best health status, while 100 points indicates the worst health status.
Body Image Assessment | At baseline and after 8 weeks
  It will be evaluated with the Multidimensional Body-Image Self-Relationship Scale (MBSRI). This scale is a scale that evaluates the body image of the individual in terms of self-attitudinal aspects. The scale also includes sub-headings that include evaluations of the individual's satisfaction with body image, physical capacity and health status. The scale consists of seven subheadings and 57 items in total. The subheadings generally provide psychological and physical evaluations. In the scale, emotional-cognitive-behavioural evaluations are made on the psychological side and physical appearance-physical competence and biological integrity evaluations are made on the physical side. A maximum score of 285 and a minimum score of 57 can be obtained from the scale.
Pulmonary Function Test (SFT) | At baseline and after 8 weeks
  In our study, SFT measurements will be performed with COSMED Pony FX device (Italy, 2011). Within the scope of the measurement rules, it will be ensured that the subjects have not eaten for at least 2 hours, have not drunk alcohol for at least 4 hours and have not smoked for at least 24 hours. In the test performed in the sitting position, the subjects will be asked to breathe normally for 4 or 5 times, then to make a deep inspiration, followed by a forced, rapid and deep expiration to release all the air. At least three repeated measurements will be performed and the measurement with the highest value in the sum of FEV1 and FVC recommended by ATS will be recorded.
Chest circumference measurement | At baseline and after 8 weeks
  It is performed to evaluate thoracic expansion, chest wall mobility and respiratory type. A bendable, non-elastic tape measure not wider than 7 mm is preferred and measurements are made with feet shoulder-width apart and body weight equally distributed on both feet. In addition, the arms should be slightly abducted for comfortable measurement. In our study, measurements will be performed from three different regions: axillary (4th costal level), epigastric (xiphoid process level) and subcostal (9th costal level) during maximal inspiration, maximal expiration and normal respiratory phase using a tape measure in standing position. The measurements will be repeated three times and the highest value will be recorded. Then, the difference between maximal inspiration and expiration will be found and recorded separately for each region.
Total body weight measurement | At baseline and after 8 weeks
  Total body weight measurement will be performed with a Tanita BC-700 (Tanita-Japan) body analyzer as weight in kilograms.
Height measurement | At baseline and after 8 weeks
  Height in meters will be measured with a height measuring tape.
Body mass index calculation | At baseline and after 8 weeks
  Weight and height will be combined to report BMI in kg/m^2).
Lower extremity fat percentage measurement | At baseline and after 8 weeks
  Lower extremity fat percentage will be measured using a Tanita BC-700 (Tanita-Japan) body analyzer.
Total body fat percentage measurement | At baseline and after 8 weeks
  Total body fat percentage measurement will be measured using a Tanita BC-700 (Tanita-Japan) body analyzer.
Lower extremity muscle percentage measurement | At baseline and after 8 weeks
  Lower extremity muscle percentage measurement will be measured using a Tanita BC-700 (Tanita-Japan) body analyzer.
Total body muscle percentage measurement | At baseline and after 8 weeks
  Total body muscle percentage measurement will be measured using a Tanita BC-700 (Tanita-Japan) body analyzer.

CONTACTS AND LOCATIONS:
Overall Officials: Onur Engin, Assist.Prof., Principal Investigator — Izmir Democracy University; Ferruh Taspinar, Prof.Dr., Principal Investigator — Izmir Democracy University
Locations (1):
- Betül TAŞPINAR, Konak, İ̇zmi̇r, Turkey (Türkiye)